CLINICAL TRIAL: NCT04998825
Title: Research on Efficacy and Tolerability of Proteoglycan F in the Treatment of Knee Osteoarthritis: a Prospective, Randomized, Double-blind Controlled Trial
Brief Title: Efficacy and Tolerability of Proteoglycan F in the Treatment of Knee Osteoarthritis
Acronym: Proteoglycan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Geriatric Hospital (Other Government)
Collaborators: Ichimaru Pharcos, Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Nguyen Trung Anh, Director, National Geriatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGH001
Record Dates: First submitted 2021-06-15; First posted 2021-08-10 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Primary Osteoarthritis of Knee Nos
Keywords: Proteoglycan F; knee osteoarthritis; Vietnam
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Prostaglandins F; Dextrins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proteoglycan F group (Experimental): * Taking Proteoglycan F
  * Dosage of Proteoglycan F: 50mg/day
  * Used time: 24 weeks
  Interventions: Dietary Supplement: Proteoglycan F
- Control group (Placebo Comparator): * Taking Placebo (Dextrin)
  * Dosage of Placebo: 50mg/day
  * Used time: 24 weeks
  Interventions: Other: Placebo product

INTERVENTIONS:
Dietary Supplement: Proteoglycan F — Salmon proteoglycan (Proteoglycan F) was extracted from salmon (Oncorhynchus keta) nasal cartilage. Salmon cartilage PG (Proteoglycan F) was manufactured in the form of a hard capsule by Ichimaru Pharcos, Co., Ltd. (at 318-1 Asagi, Motosu-shi, Gifu 501-0475 Japan) and consisted of 50 mg proteoglycan.
  Other Names: PGF
  Arms: Proteoglycan F group
Other: Placebo product — The placebo capsule contained only dextrin powder (Ichimaru Pharcos, Co., Ltd.).
  Other Names: Dextrin
  Arms: Control group

SUMMARY:
This clinical trial study is conducted in Vietnam to assess the efficacy and tolerability of Proteoglycan F in the treatment of primary knee osteoarthritis. 72 outpatients (40-80 years old) were diagnosed with primary knee osteoarthritis and met the American College of Rheumatology 1991 criteria. Patients have to be symptomatic for ≥ 3 months before enrollment and have a radiologic grade II and III measured by the Kellgren-Lawrence criteria. The study was designed as a Prospective, Randomized, Double-blind Controlled trial. Each patient will be follow during 24 weeks of intervention, follow-up every 4 weeks.

DETAILED DESCRIPTION:
With the trend of aging population and progressive increment of obesity in Vietnam, the number of patients suffering from osteoarthritis most likely will substantially increase in the coming years. Therefore, it is necessary to having a suitable and effective approach of treatment for osteoarthritis by using functional foods.

Proteoglycan is the basic substance of articular cartilage. Proteoglycans are mostly found in the extracellular matrix of animal tissue as cartilage, or in the blood vessels and brain. These substances are a key ingredient in the regeneration of cartilage, inhibiting the enzyme elastase - an intermediate that causes degenerative articular cartilage and reduces the formation of free oxygen radicals in cartilage tissue. Therefore, the effects are on inhibiting cartilage calcification, regenerating cartilage and relieving pain for cartilage degeneration, promoting cartilage metabolism, forming cartilage.

Previous studies have demonstrated that proteoglycan enhances fluid not only to alleviate arthritis pain but also prevent complications, as it gradually overcomes the damage of joint bone, resolves inflammation, helps relieve pain and prevent osteoarthritis, osteoporosis effectively. Otherwise, industrially extracted Proteoglycans presents to be safe and valuable for future studies of its function. Therefore, this randomized, double-blind controlled trial is conducted in Vietnam to assess the efficacy and tolerability of Proteoglycan F in the treatment of primary knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years old
* Diagnosed with primary knee osteoarthritis and met the American College of Rheumatology 1991 criteria
* Patients have to be symptomatic for ≥ 3 months before enrollment
* Have a radiologic grade II and III measured by the Kellgren-Lawrence criteria

Exclusion Criteria:

* Patients with secondary knee osteoarthritis
* Patients with grade-I and IV osteoarthritis (Kellgren-Lawrence)
* Patients having joint lavage, arthroscopy, or treatment with hyaluronic acid or other disease modifying agents during the previous 6 months, or treated with intra-articular corticosteroids during the past 3 months, will be excluded from the study.
* Patients have contraindications to Non-Steroidal Anti-Inflammatory Drugs
* Patients have hematologic disorders, renal disease, liver disease, diabetes mellitus, acute illness, other rheumatic diseases, disabling comorbid conditions that would make it impossible for the patient to visit the research center.
* Pregnancy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Pain relief | 6 month
  Pain intensity was assessed using the Numeric Rating Scale. Scores range from 0 to 10. The higher the score, the more severe the pain
Reduce symptoms of knee osteoarthritis 1 | 6 month
  Symptoms (pain, functionality and joints stiffness) were assessed using the Knee injury and Osteoarthritis Outcome Score. The five patient-relevant subscales of KOOS are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic assessment scales and generic measures.
Reduce symptoms of knee osteoarthritis 2 | 6 month
  Symptoms (pain, functionality and joints stiffness) were assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS), Symptoms (pain, functionality and joints stiffness) were assessed using the Lequesne index. The Lequesne index has an interview format questionnaire, including 10 questions divided into three sections regarding pain, maximum distance walked and activities of daily living. The score ranges from 0 (no pain, no disability) to 24 (maximum pain and disability)
Reduce symptoms of knee osteoarthritis 3 | 6 month
  Symptoms (pain, functionality and joints stiffness) were assessed using the Western Ontario and McMaster Universities Osteoarthritis Index. Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68)
Changes of balance, walking ability and functional mobility | 6 month
  Assessed using the Timed Up and Go test
Changes of knee joint status | 6 month
  The cartilage thickness, Joint fluid thickness, Synovial membrane thickness, was measured using knee ultrasound
The transverse relaxation time (T2) of the cartilage and Classification of other knee injuries | 6 month
  Assessed using Magnetic resonance imaging (MRI) of knee

SECONDARY OUTCOMES:
Serum cytokine levels | 6 months
  Serum cytokine levels (IL-1β, TNF-α levels)
Health related-quality of life | 6 months
  Assessed using the EuroQol 5 dimensions 5 levels questionnaires (EQ-5D-5L)

OTHER OUTCOMES:
Adverse Events | 6 months
  Any adverse events will be recorded
Liver enzymes | 6 months
  AST, ALT
Kidney function | 6 month
  ure, creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: Anh T Nguyen, PhD, Principal Investigator — National Geriatric Hospital
Locations (2):
- Vietnam (2):
  - National Geriatric Hospital, Hanoi
  - National Institution of Nutrition, Hanoi

IPD SHARING:
Plan to Share IPD: No
Will individual participant data be available (including data dictionaries)?
  * Yes
  What data in particular will be shared?
  ->Individual participant data that underlie the results reported in this article, after deidentification (text, tables,figures, and appendices).
  What other documents will be available?
  -> Study Protocol
  When will data be available (start and end dates)? --> Beginning 9 months and ending 36 months following article publication.
  With whom?
  -> Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For what types of analyses?
  -> For individual participant data meta-analysis
  By what mechanism will data be made available?
  -> Not applicable

REFERENCES:
- See also: Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the knee in osteoarthritis — https://pubmed.ncbi.nlm.nih.gov/14972335/
- See also: Evaluation of a quantitative measurement of suprapatellar effusion by ultrasonography and its association with symptoms of radiographic knee osteoarthritis: a cross-sectional observational study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4973041/
- See also: Efficacy of progressive aquatic resistance training for tibiofemoral cartilage in postmenopausal women with mild knee osteoarthritis: a randomised controlled trial — https://pubmed.ncbi.nlm.nih.gov/27211862/